CLINICAL TRIAL: NCT07348692
Title: A Phase 3, Randomized, Modified Double-blind, Active-controlled, Parallel-group, Lot-to-lot Consistency, 4-arm Study to Investigate the Safety and Immunogenicity of a 4-dose Regimen of a 21-valent Pneumococcal Conjugate Vaccine in Healthy Infants and Toddlers
Brief Title: Lot-to-lot Consistency Study of a 21-valent Pneumococcal Conjugate Vaccine in Healthy Infants From 2 Months of Age
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PSK00029; PSK00029 (Other: Sanofi Identifier); U1111-1308-6832 (Other: WHO ICTRP)
Record Dates: First submitted 2026-01-15; First posted 2026-01-16 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Pneumococcal Immunization; Healthy Volunteers
Keywords: Pneumococcal Infection; 21 Valent Pneumococcal Vaccine
MeSH Terms: conditions — Pneumococcal Infections | interventions — Vaxelis; Rotavirus Vaccines; RIX4414 vaccine; RotaTeq; Measles-Mumps-Rubella Vaccine; Chickenpox Vaccine; Hepatitis A Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants, participant's parent(s) / LAR(s), Sponsor study staff, investigators and study staff, will remain blinded during the study conduct, except dedicated study staff preparing/administering the study interventions who will be blinded regarding the PCV21 lot but unblinded regarding the patients randomized in the 20vPCV arm. The unblinded study staff will not be involved in any safety evaluation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Group 1: PCV21 (Experimental): Participants will be administered via intramuscular injection (IM) PCV21 vaccine lot 1 for Doses 1, 2 and 3; PCV21 lot 1, or different lot if needed, for Dose 4 at 2, 4, 6 and 12 months of age co-administered with routine pediatric vaccines.
  Interventions: Biological: PCV21 vaccine; Biological: Vaxelis Vaccine; Biological: Rotavirus vaccine; Biological: Measles Mumps and Rubella Vaccine; Biological: Varivax vaccine; Biological: Hepatitis A Vaccine
- Group 2: PCV21 (Experimental): Participants will be administered via IM injection PCV21 vaccine lot 2 for Doses 1, 2 and 3; PCV21 lot 2, or different lot if needed, for Dose 4 at 2, 4, 6 and 12 months of age co-administered with routine pediatric vaccines.
  Interventions: Biological: PCV21 vaccine; Biological: Vaxelis Vaccine; Biological: Rotavirus vaccine; Biological: Measles Mumps and Rubella Vaccine; Biological: Varivax vaccine; Biological: Hepatitis A Vaccine
- Group 3: PCV21 (Experimental): Participants will be administered via IM injection PCV21 vaccine lot 3 for Doses 1, 2 and 3; PCV21 lot 3, or different lot if needed, for Dose 4 at 2, 4, 6 and 12 months of age co-administered with routine pediatric vaccines.
  Interventions: Biological: PCV21 vaccine; Biological: Vaxelis Vaccine; Biological: Rotavirus vaccine; Biological: Measles Mumps and Rubella Vaccine; Biological: Varivax vaccine; Biological: Hepatitis A Vaccine
- Group 4: 20vPCV (Active Comparator): Participants will be administered via IM injection 20vPCV at 2, 4, 6 and 12 months of age co-administered with routine pediatric vaccines.
  Interventions: Biological: 20vPCV licensed vaccine; Biological: Vaxelis Vaccine; Biological: Rotavirus vaccine; Biological: Measles Mumps and Rubella Vaccine; Biological: Varivax vaccine; Biological: Hepatitis A Vaccine

INTERVENTIONS:
Biological: PCV21 vaccine — Pharmaceutical form: Suspension for injection
  Route of administration: Intramuscular
  Other Names: 515
  Arms: Group 1: PCV21; Group 2: PCV21; Group 3: PCV21
Biological: 20vPCV licensed vaccine — Pharmaceutical form: Suspension for injection
  Route of administration: Intramuscular
  Other Names: Prevnar 20™
  Arms: Group 4: 20vPCV
Biological: Vaxelis Vaccine — Pharmaceutical form: Suspension for injection
  Route of administration: Intramuscular
  Other Names: Vaxelis™
Biological: Rotavirus vaccine — Pharmaceutical form: Solution or Suspension for oral use
  Route of administration: Oral
  Other Names: Rotarix™ or RotaTeq™
Biological: Measles Mumps and Rubella Vaccine — Pharmaceutical form: Liquid solution
  Route of administration: Oral
  Other Names: M-M-R II™ or Priorix™
Biological: Varivax vaccine — Pharmaceutical form: Powder, lyophilized, for suspension for reconstitution
  Route of administration: Subcutaneous or IM
  Other Names: VARIVAX™
Biological: Hepatitis A Vaccine — Pharmaceutical form: single-dose vial or single dose prefilled syringe or suspension for injection
  Route of Administration: IM
  Other Names: VAQTA™ or Havrix™

SUMMARY:
This is a phase 3 randomized, modified double-blind study which purpose is to measure whether 3 lots of the investigational pneumococcal vaccine PCV21 can help the body to develop germ-fighting agents called "antibodies" (immunogenicity) in a similar way (ie, same immune response) when they are given in infants aged from approximately 2 months (42 to 89 days) and are safe compared to a licensed 20-valent pneumococcal vaccine (20vPCV) (Prevnar 20™).

The study duration per participant will be up to approximately 17 months. The study vaccines (either PCV21 or 20vPCV vaccines) will be administered at approximately 2, 4, 6 and 12 months of age. Routine pediatric vaccines will be given as per local recommendations.

There will be 6 study visits: Visit (V)01, V02 separated from V01 by 60 days, V03 separated from V02 by 60 days, V04 separated from V03 by 30 days, V05 at 12 months of age, V06 separated from V05 by 30 days

ELIGIBILITY:
Inclusion Criteria:

* Aged 42 to 89 days on the day of inclusion
* Participants who are healthy as determined by medical evaluation including medical history and physical examination
* Born at full term of pregnancy (≥ 37 weeks) and with a birth weight ≥ 2.5 kg or born after a gestation period above 28 (> 28 weeks) through 36 weeks with a birth weight ≥ 1.5 kg, and in both cases medically stable

Exclusion Criteria:

* Known or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy, such as anti-cancer chemotherapy or radiation therapy; or long-term systemic corticosteroid therapy
* History of microbiologically confirmed Streptococcus pneumoniae infection or disease
* Any contraindication to the routine pediatric vaccine being administered in the study
* History of seizure or significant stable or progressive neurologic disorders such as infantile spasms, inflammatory nervous system diseases, encephalopathy, cerebral palsy
* Known systemic hypersensitivity to any of the study interventions components, or history of a life-threatening reaction to the study interventions used in the study or to a product containing any of the same substances3
* Laboratory-confirmed or known thrombocytopenia, as reported by the parent(s) / legally acceptable representative (LAR(s)), contraindicating intramuscular (IM) injection.
* Bleeding disorder, or receipt of anticoagulants in the 3 weeks preceding inclusion, contraindicating IM injection.
* Chronic illness that, in the opinion of the investigator, is at a stage where it might interfere with study conduct or completion
* Moderate or severe acute illness/infection (according to investigator judgment) or febrile illness (temperature ≥ 38.0°C [≥ 100.4°F]) on the day of study intervention administration.
* Receipt of any BCG vaccine within 4 weeks preceding the first study intervention administration or planned receipt any BCG vaccine within the study period
* Previous vaccination against Streptococcus pneumoniae
* Previous vaccination against the following antigens: diphtheria, tetanus, pertussis, H. influenzae type b, poliovirus
* Receipt of more than 1 dose of hepatitis B vaccine
* Receipt of immune globulins, blood or blood-derived products since birth
* Participation at the time of study enrollment (or in the 6 weeks preceding the first study intervention administration) or planned participation during the present study period in another clinical study investigating a vaccine, drug, medical device, or medical procedure

Note: The above information is not intended to contain all considerations relevant to a potential participation in a clinical trial.

Ages: 42 Days to 89 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 896 (Estimated)
Dates: Start 2026-01-20 (Actual); Primary Completion 2028-01-19 (Estimated); Study Completion 2028-01-19 (Estimated)

PRIMARY OUTCOMES:
Serotype specific Immunoglobulin g (IgG) Geometric Mean Concentration (GMC) | 30 days after the third dose of PCV21 vaccine
  Serotype specific IgG concentrations for all serotypes included in PCV21 vaccine as measured by electrochemiluminescence assay (ECL)

SECONDARY OUTCOMES:
Serotype specific IgG concentration ≥ 0.35 µg/mL | 30 days after the third dose of PCV21 vaccine
  Serotype specific IgG concentration ≥ 0.35 μg/mL (seroresponse) for all serotypes included in PCV21 as measured by ECL
Presence of any immediate adverse events (AEs) | Within 30 minutes after each vaccine injection
  Number of participants experiencing immediate AEs
Presence of solicited injection site and systemic reactions through 7 days after each vaccine injection | Through 7 days after each vaccine injection
  Number of participants experiencing solicited injection site and systemic reactions
Presence of unsolicited (spontaneously reported) injection site reactions and unsolicited systemic AEs | Through 30 days after each vaccine injection
  Number of participants experiencing unsolicited injection site reactions and unsolicited systemic AEs
Presence of serious adverse events (SAEs) and adverse events of special interest (AESIs) throughout the study | Throughout the study (through 6 months post-last vaccine injection)
  Number of participants experiencing SAEs and AESIs

CONTACTS AND LOCATIONS:
Locations (3):
- Honduras (3):
  - Investigational Site Number : 3400001, San Pedro Sula
  - Investigational Site Number : 3400002, Tegucigalpa
  - Investigational Site Number : 3400003, Tegucigalpa

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org